CLINICAL TRIAL: NCT07378800
Title: Fostering Positive Care Interactions in Assisted Living
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Rachel McPherson, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AARG-25-1481519
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Dementia
Keywords: positive care interactions
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FPCI-AL (Experimental): The FPCI-AL is implemented using a research facilitator working with a community-based champion and stakeholder group to provide the following four-steps: (1) assessments of the environment and policy to facilitate positive interactions; (2) educating staff on fostering positive interactions; (3) establishing individualized positive care interaction approaches for residents and incorporating them into resident service plans; and (4) providing ongoing mentoring, motivating, and role modeling for staff to reinforce positive care interactions.
  Interventions: Behavioral: FPCI-AL
- Education Only (EO) (Active Comparator): Communities randomized to education only will receive the same education as provided in FPCI-AL step two via an established PowerPoint. Delivery format will match community preferences (e.g., online or in-person) for pragmatic reasons and to facilitate the education process.
  Interventions: Behavioral: Education Only (EO)

INTERVENTIONS:
Behavioral: FPCI-AL — Following randomization, champions and stakeholder team members from the communities will be identified. The investigators will recommend the following individuals to be members of the stakeholder team: assisted living administrator, nurse manager, nursing assistant, and activity and rehabilitation staff as available.
  Following the initial team meeting, the research facilitator will work with each treatment assisted living community for eight hours weekly during months one and two, and then for four hours weekly for the remaining four months using a face-to-face approach to implement the four components of the FPCI-AL.
  Arms: FPCI-AL
Behavioral: Education Only (EO) — Communities randomized to education only will receive the same education as provided in FPCI-AL step two via an established PowerPoint. Delivery format will match community preferences (e.g., online or in-person) for pragmatic reasons and to facilitate the education process.
  Arms: Education Only (EO)

SUMMARY:
The purpose of this study is to improve the quality of staff-resident care interactions particularly among residents living with Alzheimer's disease or related dementias (ADRD ) by testing the Fostering Positive Care Interactions in Assisted Living (FPCI-AL) intervention. This study will be a critical first step in determining the sample size needed to test the efficacy of a practical approach to improving the quality of care interactions for assisted living residents living with ADRD, ultimately enhancing behavioral outcomes such as decreasing behavioral symptoms of distress, reducing resistiveness to care, and optimizing engagement in care tasks.

DETAILED DESCRIPTION:
Staff-resident care interactions are integral to effective care provision in assisted living communities, and especially critical for residents living Alzheimer's disease or related dementias (ADRD). The purpose of this study is to improve the quality of staff-resident care interactions particularly among residents living with ADRD by testing the Fostering Positive Care Interactions in Assisted Living (FPCI-AL) intervention. This 6 month intervention uses a four-step, theoretically based approach implemented by a research facilitator to change how staff provide care to residents living with ADRD. The research facilitator will work with a community-based stakeholder team and identified champion to implement the following four-step approach: 1) assessments of the environment and policy to facilitate positive interactions; (2) educating staff on fostering positive interactions; (3) establishing individualized positive care interaction approaches for residents and incorporating them into resident service plans; and (4) providing ongoing mentoring, motivating, and role modeling for staff to reinforce positive care interactions. Therefore, the aims of this study are to: Aim 1: Establish the feasibility of the FPCI-AL based on delivery, receipt and enactment of study activities; and establish acceptability of the FPCI-AL; Aim 2: Evaluate the preliminary efficacy of the FPCI-AL on the quality of care interactions received by residents living with ADRD; and Aim 3: Evaluate the preliminary efficacy of the FPCI-AL on behavioral symptoms of distress, resistiveness to care, and resident engagement with staff during care interactions. The investigators will use a cluster randomized controlled trial with a repeated measures design to test the feasibility and preliminary efficacy of the FPCI-AL. This study will include four assisted living communities, and a convenience sample of 25 residents per community (N = 100) will be recruited. Residents will be eligible to participate if they: (a) are 55 years of age or older; (b) are currently residing in a participating community; and (c) have evidence of ADRD based on a score ≤20 on the Saint Louis University Mental Status Examination. Residents will be excluded if they are admitted to the assisted living for short term care. The research facilitator will implement the four intervention steps over 6 months. Communities randomized to Education Only will receive education consistent with step two of the FPCI-AL. All community and resident data will be obtained by a trained research evaluator and will be measured at baseline, 4 months, and 6 months post-intervention. This study will be a critical first step in determining the sample size needed to test the efficacy of a practical approach to improving the quality of care interactions for assisted living residents living with ADRD, ultimately enhancing behavioral outcomes such as decreasing behavioral symptoms of distress, reducing resistiveness to care, and optimizing engagement in care tasks.

ELIGIBILITY:
Inclusion Criteria:

* 55 years of age or older
* currently residing in a participating community
* Evidence of ADRD based on a score ≤20 on the Saint Louis University Mental Status Examination

Exclusion Criteria:

* Admitted to the assisted living for short term care

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Modified Quality of Interactions Scale | Baseline, 4 months, 6 months
  Quality of care interactions will be measured using the Modified Quality of Interactions Scale, an observational tool that measures interaction characteristics and quality using a quantified scoring system. It records the care interaction location, type of care activity, and type of care provider in care (e.g., nurse). The total score ranges from 0 to 7, with higher scores indicating better, more positive interactions.

SECONDARY OUTCOMES:
Neuropsychiatric Inventory Questionnaire | Baseline, 4 months, 6 months
  The Neuropsychiatric Inventory Questionnaire (NPI-Q) assesses the presence, severity, and impact on caregivers of 12 behavioral symptoms of distress (e.g., delusions, hallucinations, anxiety). For the purposes of this study only the presence of behavior will be considered. The total score ranges from 0 to 12, with higher numbers indicating more behavioral symptoms of distress.
Resistiveness to Care Scale | Baseline, 4 months, 6 months
  Resistiveness to care will be assessed during care interactions using the Resistiveness to Care Scale, which measures the frequency of 16 resistive behaviors (e.g., kicking, hitting). The total score ranges from 0 to 16, with higher scores indicating more resistiveness to care behaviors.
Resident Engagement with Staff During Care Interactions | Baseline, 4 months, 6 months
  The Modified Quality of Interaction Scale item, "What is the level of resident engagement?", will be used during assessments of staff-resident care interactions to record resident engagement as active, passive, or restrictive.

IPD SHARING:
Plan to Share IPD: No